CLINICAL TRIAL: NCT02859779
Title: Needs Assessment of Mediterranean Adolescents With Type 1 Diabetes About Therapeutic Education Sessions: A Qualitative Study
Brief Title: Needs Assessment of Mediterranean Adolescents With Type 1 Diabetes About Therapeutic Education Sessions
Acronym: BADET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-36
Record Dates: First submitted 2016-08-01; First posted 2016-08-09 (Estimated); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Type 1 Diabetes in Adolescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mediterranean adolescents with type 1 diabetes (Other)
  Interventions: Behavioral: education programs

INTERVENTIONS:
Behavioral: education programs — Four audio-recorded discussion groups will be organized in each of the 10 clinical settings

SUMMARY:
Background: In type 1 diabetes, adolescence is often associated with deterioration in glycemic control, attributed to a poorly monitored diet, little exercise, poor treatment compliance, risk behaviors, endocrine changes with puberty, leading to greater resistance to insulin. Therapeutic patient education (TPE) is the key to successful management of the disease and treatment for adolescents with type 1 diabetes. Ten TPE programs exist in the Mediterranean region in France, and the care teams implementing them wish to promote joint reflection with sick teenagers and families to identify needs and expectations of everyone on priority skills to develop, to promote better management of the disease and improved quality of life.

Aim: To study the needs and expectations of adolescents with type 1 diabetes for skills to be developed during the educational sessions, to promote self-management of their disease and their treatment.

Method: Four audio-recorded focus groups will be organized in all 10 clinical settings (adolescents, parents and health professionals). Thematic analysis will be carried out from the transcript of the focus groups.

Expected results: The results will allow a joint reflection involving the participation of young patients, families, health professionals and the research team to build and implement new educational sessions that meet the identified needs. This action resulting from the research is expected to pool resources in different health facilities providing therapeutic education programs and to harmonize practices.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 11 and 16 years inclusive
* Type 1 diabetes diagnosis confirmed by a physician according to the diagnostic criteria
* Monitoring in the institutions participating in the research
* Speaking the French language (elementary level)
* Consent signed by the holders of the exercise of parental authority and the participant

Exclusion Criteria:

* Pregnant women, parturient women or breastfeeding mothers
* Persons deprived of liberty by a judicial or administrative decision
* Those hospitalized without consent under articles L. 3212-1 and L. 3213-1 that do not fall under the provisions of Article L. 1121-8
* Persons admitted in a health or social institution for purposes other than research (art. L.1121-6 health public code)

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-02-04 (Actual); Primary Completion 2017-04-12 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Needs and expectations of adolescents with type 1 diabetes for skills to be developed during the educational sessions | one day
  An interview guide was developed from the regulatory framework of therapeutic education in France, the theoretical framework of psychosocial skills in social psychology of health and from a previous experiment in the UK with diabetic children and their parents, to develop communication skills of health professionals (Hawthorne et al., 2011)

SECONDARY OUTCOMES:
Needs and expectations of parents of adolescents with type 1 diabetes for skills to be developed during the educational sessions | one day
  An interview guide was developed from the regulatory framework of therapeutic education in France, the theoretical framework of psychosocial skills in social psychology of health and from a previous experiment in the UK with diabetic children and their parents, to develop communication skills of health professionals (Hawthorne et al., 2011)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Timone Assistance Publique Hôpitaux de Marseille, Marseille, France